CLINICAL TRIAL: NCT06978101
Title: Correlation Between Visual Field Changes and OCT Angiographic Chorioretinal Changes in Patients With Primary Open Angle Glaucoma
Brief Title: Visual Field Changes and OCT Angiographic Chorioretinal Changes in Patients With Primary Open Angle Glaucoma
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Miadaa Hassan Hassaneen, Assistant Lecturer of Ophthalmology Department, Al-Azhar Faculty of Medicine in Assiut., Assiut University
Other Study IDs: MD/AZ.AST./OPH026/10/191/1/202
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Visual Field; OCT Angiography; Chorioretinal Changes; Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POAG group: Patients had intraocular pressure (IOP)>21 mmHg,
  Interventions: Other: POAG group
- Control group: Patients without family history of primary open-angle glaucoma (POAG), IOP ˂21mm Hg.
  Interventions: Other: Control group

INTERVENTIONS:
Other: POAG group — Patients had intraocular pressure (IOP)>21 mmHg.
  Groups: POAG group
Other: Control group — Patients without family history of primary open-angle glaucoma (POAG), IOP ˂21mm Hg.
  Groups: Control group

SUMMARY:
This study aimed to assess the correlation between visual field changes and optical coherence tomography (OCT) angiography changes of retinal nerve fiber layer in patients with primary open angle glaucoma.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide. Since glaucomatous damage is preventable but irreversible, an early diagnosis and close follow-up of glaucoma patients are primordial. Optical coherence tomography angiography (OCTA) is a recently developed, noninvasive imaging modality that detects blood flow through the motion contrast generated by red blood cells.

Currently, there are 2 groups of complementary exams used for the diagnosis and follow-up of glaucoma patients: structural (where OCT has a considerable role) and functional (visual field) optic nerve measurements, Both technologies have strengths and limitations.

A new technology for diagnosis and follow-up that can avoid the limitations summarized above is lacking. OCTA seems to be a good candidate for such a role, OCT can detect the Doppler frequency shift of the backscattered light that provides information on blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma patients.

Exclusion Criteria:

1. Hazy media.
2. Diabetic Retinopathy.
3. Uveitis.
4. Other Glaucomas

   * Acute congestive glaucoma
   * Secondary glaucomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort nonrandomized trial was carried out on 100 cases with primary open-angle glaucoma (POAG) group (n=80): had intraocular pressure (IOP)>21 mmHg, and control group (n=20): without family history of POAG, IOP ˂21mm Hg.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Peripapillary vessel density (PpVD) | 12 months post-procedure
  Peripapillary vessel density (PpVD) was examined with swept-source OCT(DRI OCT Triton;Topcon Corporation,Tokyo,Japan) after pupillary dilatation , using an optic disc scan , peripapillary vessel density was derived from the images acquired with a 6 mm x6 mm mm field of view centered on the optic disc.
  PpVD measurements were calculated within the RNFL in a slab from the internal limiting membrane (ILM) to the RNFL posterior boundary.

SECONDARY OUTCOMES:
Pattern standard deviation (PSD) | 12 months post-procedure
  Pattern standard deviation ( PSD) on Visual field test was performed with the Swedish Interactive Threshold Algorithm (SITA) Standard strategy program 24-2 of the octopus polar analysis which measures 24 degrees temporally and 30 degrees nasally and test 54 points.
Mean deviation (MD) | 12 months post-procedure
  Mean deviation(MD) on Visual field test was performed with the Swedish Interactive Threshold Algorithm (SITA) Standard strategy program 24-2 of the octopus polar analysis which measures 24 degrees temporally and 30 degrees nasally and test 54 points.
The thickness of the peripapillary retinal nerve fiber layer(RNFL) | 12 months post-procedure
  The thickness of the peripapillary retinal nerve fiber layer(RNFL) was obtained from a circle with a diameter of 3.4 mm centered on the optic disc.
  The RNFL thickness in 4 quadrants and 12 clock-hour were obtained by using the built-in automated segmentation algorism of the system.
Intraocular pressure (IOP) | 12 months post-procedure
  Intraocular pressure (IOP) was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author